CLINICAL TRIAL: NCT06168539
Title: Reduction of Microemboli of Air Using a New Developed Air Trap (EmbolessTM) During Haemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CIV-20-02-031667
Record Dates: First submitted 2023-11-06; First posted 2023-12-13 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-01

CONDITIONS: Hemodialysis Complication; Air Embolism; Extracorporeal Circulation; Complications
MeSH Terms: conditions — Embolism, Air

STUDY DESIGN:
Intervention Model Description: Each patient is randomized to start with either standard or intervention vice versa. Paired analyses are done.
Masking Description: Measuring data of microemboli counts is masked for the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (Active Comparator): A regular standard dialysis is performed and held as active comparator for analysis
  Interventions: Other: Standard
- Emboless (Experimental): Emboless tubing set is part of the extracorporeal venous bloodline instead of the venous chamber by Fresenius (see standard above).
  For more information see reference Jonsson et al 2023- mentioned in references.
  Interventions: Other: Emboless

INTERVENTIONS:
Other: Emboless — Emboless has the US patent number 8894749 is compared to standard dialysis See also reference Jonsson et al 2023 referred to in the main text.
  Arms: Emboless
Other: Standard — Standard dialysis set is used as comparative
  Arms: Standard

SUMMARY:
During hemodialysis (HD) the blood of the patient pass an extracorporeal circuit that contains a dialyzer for rinsing and a venous chamber (air trap) to prevent from air embolism through the return blood into the patient. However, air traps in clinical use have limited capacity to prevent from microemboli of air to enter the return bloodline and deposit as emboli in the body such as lungs, heart and brain. The Investigator developed the air trap Emboless that was patented. In vitro studies showed significantly better reduction of microemboli contaminations than air traps compared to that in clinical use.

The present randomized clinical trial compares two different air traps used by the same patients in a cross-over design (as pairs) using the Emboless compared with the Fresenius 4008/5008 (F5008).

Chronic HD patients are randomized to perform the first HD with either their standard air trap (F5008) in the venous bloodline tubing or using the Emboless bloodline and vice versa. Each patient was included to make two paired series. A safety committee evaluates if significantly worse outcome appears especially with the Emboless, to stop the study.

During HD the microbubbles are counted by a GAMPT ultrasound device using two probes. One probe is set at the inlet side of the air trap and the second at the outlet side. The outlet side represents data of microbubbles in the blood that are entering into the patient. Comparative non-parametric paired analyses are performed between the air traps.

Monitoring of the study is performed.

DETAILED DESCRIPTION:
During hemodialysis (HD) the blood of the patient pass an extracorporeal circuit that contains a dialyzer for rinsing and a venous chamber (air trap) to prevent from air embolism through the return blood into the patient. However, air traps in clinical use have limited capacity to prevent from microemboli of air to enter the return bloodline and deposit as emboli in the body such as lungs, heart and brain. The Investigator developed the air trap Emboless that was patented in Europe, USA and India. In vitro studies showed significantly better reduction of microemboli contaminations than air traps compared to that in clinical use.

The present randomized clinical trial compares two different air traps used by the same patients in a cross-over design (as pairs) using the Emboless compared with the Fresenius 4008/5008 (F5008).

Chronic HD patients are randomized to perform the first HD with either their standard air trap (F5008) in the venous bloodline tubing or using the Emboless bloodline and vice versa. Each patient is included to make two paired series. A maximum of 30 patients are planned. Each with 2 series of each two different sets of air traps that would give a total of 120 dialyses. A safety committee evaluates if significantly worse outcome appears especially with the Emboless.

During HD the microbubbles are counted by a GAMPT ultrasound device using two probes. One probe is set at the inlet side of the air trap and the second at the outlet side. The outlet side represents data of microbubbles in the blood that are entering into the patient. Comparative non-parametric paired analyses are performed between the air traps.

Monitoring of the study is performed.

ELIGIBILITY:
Inclusion Criteria:

Accepted are all patients performing chronic HD due to End Stage renal disease of any reason:

* 18 years and older
* accept, by consent, to participate in the study
* both genders,
* any ethnicity

Exclusion Criteria:

Patients that are expected not to fulfil a whole series of two dialysis within the study such as those:

* who suffer from active cancer or severe infection, cachexia or are planned for kidney transplantation close to the study period.
* patients that by any reason are considered inappropriate by the principal investigator, such as patients that experience severe hypotensive episodes during standard dialysis.

Home-haemodialysis treatments and self-care dialysis treatments are not included in the study. If such patient accepts to participate in the study, he/she has to adapt to study criteria (assisted treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — consecutively based on the approval of patients. Excluding those with active infections.
Enrollment: 20 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Comparison of change in air micro bubbles during hemodialysis | 1 year
  Numbers of air micro bubbles (diameter sizes from 20-500µm diameter) are counted at inlet and outlet of the air trap with parallel probes using ultrasound GAMPT 200 device during 30minutes of HD. A calculation clarifies change in percentage of outlet versus inlet amount/size of microbubble air return into the return bloodline that is connected to the return needle placed in the vein of the patient. The size in diameter and numbers within the dialysis time/30 minutes of HD are given.

SECONDARY OUTCOMES:
Comparison of change in air micro bubbles for hemodialysis versus hemodiafiltration | 1 year
  The Investigator aims to compare the microbubble reduction of the air traps also between the hemodialysis versus hemodiafiltration if the specific patient performs this dialysis under normal circumstances.
adverse events | 1 year
  If a patient experience adverse events these will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Forsberg, MD, PhD, Principal Investigator — Region Vasterbotten Skelleftea Hospital, Sweden
Locations (1):
- Region Vasterbotten, Skelleftea Sjukhus, Dialysen, Skellefteå, Sweden

IPD SHARING:
Plan to Share IPD: Yes
We can share data upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Expected time of completing data is 1 year from now.
Access Criteria: Reasonable request to share information such as safety analyses, repeating studies or control authorities.

REFERENCES:
- [Background] Stegmayr BG. Sources of Mortality on Dialysis with an Emphasis on Microemboli. Semin Dial. 2016 Nov;29(6):442-446. doi: 10.1111/sdi.12527. Epub 2016 Aug 16. PMID 27528100
- [Background] Stegmayr B. Air contamination during hemodialysis should be minimized. Hemodial Int. 2017 Apr;21(2):168-172. doi: 10.1111/hdi.12474. Epub 2016 Aug 30. PMID 27576675
- [Background] Matsuda K, Fissell R, Ash S, Stegmayr B. Long-Term Survival for Hemodialysis Patients Differ in Japan Versus Europe and the USA. What Might the Reasons Be? Artif Organs. 2018 Dec;42(12):1112-1118. doi: 10.1111/aor.13363. Epub 2018 Nov 11. No abstract available. PMID 30417399
- [Result] Forsberg U, Jonsson P, Stegmayr B. Air contamination during medical treatment results in deposits of microemboli in the lungs: An autopsy study. Int J Artif Organs. 2019 Sep;42(9):477-481. doi: 10.1177/0391398819840363. Epub 2019 Apr 11. PMID 30973284
- [Result] Forsberg U, Jonsson P, Stegmayr B. Microemboli induced by air bubbles may be deposited in organs as a consequence of contamination during medical care. Clin Kidney J. 2022 Oct 6;16(1):159-166. doi: 10.1093/ckj/sfac217. eCollection 2023 Jan. PMID 36726427
- [Result] Jonsson P, Stegmayr C, Stegmayr B, Forsberg U. Venous chambers in clinical use for hemodialysis have limited capacity to eliminate microbubbles from entering the return bloodline: An in vitro study. Artif Organs. 2023 Jun;47(6):961-970. doi: 10.1111/aor.14495. Epub 2023 Jan 10. PMID 36594759